CLINICAL TRIAL: NCT01637922
Title: Effect of Multiple Dosing With BI 201335 on the Safety, Pharmacokinetics and Pharmacodynamics of Steady-state Methadone and Buprenorphine/Naloxone in Subjects on Stable Addiction Management Therapy
Brief Title: Drug Interaction Study With BI 201335 and Methadone or Buprenorphine/Naloxone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1220.57
Record Dates: First submitted 2012-07-09; First posted 2012-07-11 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2015-07

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — faldaprevir

ARMS (2):
- Methadone group (Active Comparator): patients on stable methadone therapy (at least 30 days) up to a maximum of 180mg per day
  Interventions: Drug: BI 201335
- Buprenorphine (Active Comparator): patients on stable buprenorphine/naloxone therapy (at least 30 days) up to a maximum dose of 24mg/6mg per day.
  Interventions: Drug: BI 201335

INTERVENTIONS:
Drug: BI 201335 — BI 201335 for 9 days
  Arms: Methadone group
Drug: BI 201335 — BI 201335 for 9 days
  Arms: Buprenorphine

SUMMARY:
Otherwise healthy subjects who are currently bein maintained on either methadone or buprenorphine/naloxone for opioid maintenance therapy who have been on a stable dose for at least 30 days will be administered BI 201335 daily to determine if a drug interaction occurs between BI 201335 and either methadone or buprenorphine/naloxone.

ELIGIBILITY:
Inclusion criteria:

1. stable dose of either methadone or buprenorphine/naloxone for 30 days for opioid maintenance therapy.
2. Male and female volunteers with a body mass index (BMI) = 18.5 and < 32 with a minimum weight of 50kg.

Exclusion criteria:

1. any other significant medical illness of clinical significance.
2. history of rash or photosensitivity
3. chronic or acute infections including HIV, hepatitis B and hepatitis C.
4. history of allergy considered significant for this study
5. intake of any other medications except for methadone or buprenorphine/naloxone.
6. QTc on electrocardiogram (ECG) > 470.
7. use of any other investigational drug within 30 days of the study.
8. drug or alcohol abuse (other than the defined opioid maintenance therapy with either methadone or buprenorphine/naloxone)
9. blood donation of more than 100mL within four weeks of the trial.
10. excessive physical activities one week prior to and during the trial.
11. any clinically relevant laboratory value.
12. concomitant use of any food product known to alter P450 or P-gp activity such as grapefruit juice, seville oranges and St. John's Wort.
13. inadequate venous access

    For women of childbearing potential:
14. pregnancy or planning to become pregnant within 3 months of the trial
15. positive pregnancy test at screening visit
16. no proof of sterilization or unwilling or unable to use a double barrier method of birth control during the study and up to 3 months after the study.
17. lactation with active breastfeeding from screening up to 30 days after last study visit.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- United States (3):
  - 1220.57.0001 Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - 1220.57.0002 Boehringer Ingelheim Investigational Site, Overland Park, Kansas
  - 1220.57.0003 Boehringer Ingelheim Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Joseph D, Schobelock MJ, Riesenberg RR, Vince BD, Webster LR, Adeniji A, Elgadi M, Huang F. Effect of steady-state faldaprevir on the pharmacokinetics of steady-state methadone and buprenorphine-naloxone in subjects receiving stable addiction management therapy. Antimicrob Agents Chemother. 2015 Jan;59(1):498-504. doi: 10.1128/AAC.04046-14. Epub 2014 Nov 10. PMID 25385094

RESULTS

PARTICIPANT FLOW:
Groups:
- Methadone Group: patients on stable methadone therapy (at least 30 days) up to a maximum of 180mg per day. Days 1-13.
  BI 201335(faldaprevir): Oral dose of BI 201335(faldaprevir) 480 mg on day 2 and 240 mg twice daily for days 3 to 9.
- Buprenorphine/Naloxone (Suboxone): patients on stable buprenorphine/naloxone therapy (at least 30 days) up to a maximum dose of 24mg/6mg per day. Days 1-13.
  BI 201335(faldaprevir): Oral dose of BI 201335(faldaprevir) 480 mg on day 2 and 240 mg twice daily for days 3 to 9.
Period: Overall Study
Arm/Group | Methadone Group | Buprenorphine/Naloxone (Suboxone)
Started | 15 | 19
Completed | 13 | 14
Not Completed | 2 | 5
Not completed — Adverse Event | 0 | 1
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: This set included all subjects who were dispensed study medication and were documented to have taken at least one dose of study drug.
Groups:
- Methadone Group: patients on stable methadone therapy (at least 30 days) up to a maximum of 180mg per day. Days 1-13.
  BI 201335(faldaprevir): BI 201335(faldaprevir) for days 3 to 9.
- Buprenorphine/Naloxone (Suboxone): patients on stable buprenorphine/naloxone therapy (at least 30 days) up to a maximum dose of 24mg/6mg per day. Days 1-13.
  BI 201335(faldaprevir): BI 201335(faldaprevir) for days 3 to 9.
- Total: Total of all reporting groups
Arm/Group | Methadone Group | Buprenorphine/Naloxone (Suboxone) | Total
Number analyzed (Participants) | 15 | 19 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.4 (11.0) | 34.1 (8.7) | 34.6 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 11 | 16 | 27

OUTCOME MEASURES:

1. Primary Outcome: R-methadone: Geometric Mean Steady-state AUC0-24 on Day 1 and on Day 9.
Description: These are the unadjusted summary statistics on the original scale for area under the concentration time curve (AUC) of faldaprevir in plasma over a uniform dosing interval from 0 to 24 hours.
Time Frame: 0 hours, 0.5 hours, 1 hour, 1.5 hours, 2 hours, 2.5 hours, 3 hours, 4 hours, 6 hours, 8 hours, 12 hours and 24 hours on Day 1 and Day 9
Population: This set included all subjects who took at least one dose of study drug and had evaluable data for at least one observation for at least one primary endpoint. Subjects considered to be not evaluable, if the subject had a protocol deviation relevant to relative bioavailability. Or experienced emesis and vomiting at or before two times median tmax.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng*h/mL]
Arm/Group | Methadone Group
Number analyzed (Participants) | 15
[ng*h/mL]
  R-methadone with FDV (Day 9) | 6990 (31.7)
  R-methadone alone (Day 1) | 5920 (37.2)
Statistical Analysis 1: Comparison: Methadone Group; Methadone(MTD) + Faldaprevir(FDV) on Day 9 vs. Methadone(MTD) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.1638, ANOVA — p-value for ratio outside interval 80% to 125%; Log transformed endpoints were analyzed using an ANOVA model, including treatment as a fixed effect and subject as a random effect; Geometric mean ratio (%) = 118.12, 90% CI 2-sided [107.06 to 130.32], Standard Deviation 15.4 — The standard deviation is actually the intra-individual geometric coefficient of variation

2. Primary Outcome: R-methadone: Geometric Mean Steady-state Cmax on Day 1 and on Day 9.
Description: These are the unadjusted summary statistics on the original scale for the maximum measured concentration of faldaprevir in plasma at steady state.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng/ml]
Arm/Group | Methadone Group
Number analyzed (Participants) | 15
[ng/ml]
  R-methadone with FDV (Day 9) | 393 (29.8)
  R-methadone alone (Day 1) | 345 (33.3)
Statistical Analysis 1: Comparison: Methadone Group; Methadone(MTD) + Faldaprevir(FDV) on Day 9 vs. Methadone(MTD) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0391, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 114.08, 90% CI 2-sided [104.812 to 124.164], Standard Deviation 13.2 — The standard deviation is actually the intra-individual geometric coefficient of variation

3. Primary Outcome: R-methadone: Geometric Mean Steady-state C24hr on Day 1 and on Day 9.
Description: These are the unadjusted summary statistics on the original scale for steady-state plasma concentration of faldaprevir 24 hours after the last dose
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng/mL]
Arm/Group | Methadone Group
Number analyzed (Participants) | 15
[ng/mL]
  R-methadone with FDV (Day 9) | 235 (36.8)
  R-methadone alone (Day 1) | 210 (39.4)
Statistical Analysis 1: Comparison: Methadone Group; Methadone(MTD) + Faldaprevir(FDV) on Day 9 vs. Methadone(MTD) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0603, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 111.79, 90% CI 2-sided [99.243 to 125.922], Standard Deviation 18.7 — The standard deviation is actually the intra-individual geometric coefficient of variation

4. Primary Outcome: S-methadone: Geometric Mean Steady-state AUC0-24 on Day 1 and on Day 9
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng*h/ml]
Arm/Group | Methadone Group
Number analyzed (Participants) | 15
[ng*h/ml]
  S-methadone with FDV (Day 9) | 7610 (39.3)
  S-methadone alone (Day 1) | 6470 (41.5)
Statistical Analysis 1: Comparison: Methadone Group; S-Methadone(MTD) + Faldaprevir(FDV) on Day 9 vs. S-Methadone(MTD) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.1424, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 117.65, 90% CI 2-sided [106.89 to 129.50], Standard Deviation 15.0 — The standard deviation is actually the intra-individual geometric coefficient of variation

5. Primary Outcome: S-methadone: Geometric Mean Steady-state Cmax on Day 1 and on Day 9
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng/mL]
Arm/Group | Methadone Group
Number analyzed (Participants) | 15
[ng/mL]
  S-methadone with FDV (Day 9) | 474 (36.6)
  S-methadone alone (Day 1) | 425 (34.9)
Statistical Analysis 1: Comparison: Methadone Group; S-Methadone(MTD) + Faldaprevir(FDV) on Day 9 vs. S-Methadone(MTD) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0367, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 111.46, 90% CI 2-sided [100.420 to 123.715], Standard Deviation 16.3 — The standard deviation is actually the intra-individual geometric coefficient of variation

6. Primary Outcome: S-methadone: Geometric Mean Steady-state C24hr on Day 1 and on Day 9
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [ng/mL]
Arm/Group | Methadone Group
Number analyzed (Participants) | 15
[ng/mL]
  S-methadone with FDV (Day 9) | 231 (46.3)
  S-methadone alone (Day 1) | 207 (48.8)
Statistical Analysis 1: Comparison: Methadone Group; S-Methadone(MTD) + Faldaprevir(FDV) on Day 9 vs. S-Methadone(MTD) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0488, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 111.52, 90% CI 2-sided [99.577 to 124.888], Standard Deviation 17.7 — The standard deviation is actually the intra-individual geometric coefficient of variation

7. Secondary Outcome: Pharmacodynamic Assessment of Withdrawal From Either Methadone or Buprenorphine/Naloxone Using the Objective Opiate Withdrawal Scale (OOWS)-Change From Baseline
Description: The OOWS is conducted by a trained independent examiner for either the presence or absence of the following symptoms during a 10 minute observation period at designated times during the trial. The minimum possible OOWS score is 0 and the maximum possible score is 13. Objective criteria: Yawning, Rhinorrhoea, Piloerection, perspiration, lacrimation, mydriasis, hot and cold flushes, restlessness, vomiting, tremors, anxiety, muscle twitches, abdominal cramps. Higher score indicates increasing severity of opiate withdrawal syndrome.
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12 and End of treatment
Population: This set included all subjects who took at least one dose of study drug.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Methadone Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 15 | 19
units on a scale
  Day 2 | 0.0 [-1 to 1] | 0.0 [-2 to 1]
  Day 3 | 0.0 [-1 to 1] | 0.0 [-2 to 1]
  Day 4 (N=15,18) | 0.0 [-2 to 1] | 0.0 [-3 to 1]
  Day 5 (N=15,18) | 0.0 [-1 to 0] | 0.0 [-3 to 1]
  Day 6 (N=15,18) | 0.0 [-1 to 0] | 0.0 [-3 to 2]
  Day 7 (N=15,15) | 0.0 [-1 to 1] | 0.0 [-2 to 1]
  Day 8 (N=15,15) | 0.0 [-1 to 0] | 0.0 [-3 to 1]
  Day 9 (N=15,15) | 0.0 [-1 to 1] | 0.0 [-2 to 2]
  Day 10 (N=15,15) | 0.0 [-1 to 1] | 0.0 [-2 to 1]
  Day 11 (N=15,15) | 0.0 [-1 to 1] | 0.0 [-3 to 0]
  Day 12 (N=15,15) | 0.0 [-1 to 1] | 0.0 [-3 to 1]
  End of Treatment (EOT) (N=14,16) | 0.0 [-1 to 2] | 0.0 [-3 to 1]
Statistical Analysis 1: Comparison: Methadone Group; Pearson correlation of trough concentrations of R-methadone and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.01098, 95% CI 2-sided [-0.189801 to 0.168640]
Statistical Analysis 2: Comparison: Methadone Group; Pearson correlation of change from baseline for trough concentrations of R-methadone and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.10188, 95% CI 2-sided [-0.287471 to 0.092062]
Statistical Analysis 3: Comparison: Methadone Group; Pearson correlation of trough concentrations of S-methadone and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.03198, 95% CI 2-sided [-0.209893 to 0.148238]
Statistical Analysis 4: Comparison: Methadone Group; Pearson correlation of change from baseline for trough concentrations of S-methadone and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.00260, 95% CI 2-sided [-0.189172 to 0.194156]
Statistical Analysis 5: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of trough concentrations of Buprenorphine and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.03364, 95% CI 2-sided [-0.214505 to 0.149733]
Statistical Analysis 6: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of change from baseline for trough concentrations of Buprenorphine and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.14703, 95% CI 2-sided [-0.404929 to 0.135425]
Statistical Analysis 7: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of trough concentrations of norbuprenorphine and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.05431, 95% CI 2-sided [-0.240578 to 0.136305]
Statistical Analysis 8: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of change from baseline for trough concentrations of norbuprenorphine and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.09727, 95% CI 2-sided [-0.344024 to 0.163687]
Statistical Analysis 9: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of trough concentrations of naloxone and OOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.36105 — Confidence interval is not provided due to sparse data. There was only 1 patient for this analysis

8. Primary Outcome: Buprenorphine: Geometric Mean Steady-state AUC0-24 on Day 1 and on Day 9.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg*h/ml]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 13
[pg*h/ml]
  BUPRENORPHINE with FDV (Day 9) | 58700 (73.1)
  BUPRENORPHINE alone (Day 1) | 54000 (86.5)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); BUPRENORPHINE(BUP) + Faldaprevir(FDV) on Day 9 vs. BUPRENORPHINE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.1642, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 108.71, 90% CI 2-sided [85.14 to 138.80], Standard Deviation 36.1 — The standard deviation is actually the intra-individual geometric coefficient of variation

9. Primary Outcome: Buprenorphine: Geometric Mean Steady-state Cmax on Day 1 and on Day 9.
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg/ml]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 13
[pg/ml]
  BUPRENORPHINE with FDV (Day 9) | 7610 (74.5)
  BUPRENORPHINE alone (Day 1) | 8240 (92.0)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); BUPRENORPHINE(BUP) + Faldaprevir(FDV) on Day 9 vs. BUPRENORPHINE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.1420, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 92.43, 90% CI 2-sided [73.48 to 116.27], Standard Deviation 33.7 — The standard deviation is actually the intra-individual geometric coefficient of variation

10. Primary Outcome: Buprenorphine: Geometric Mean Steady-state C24hr on Day 1 and on Day 9.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg/mL]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 12
[pg/mL]
  BUPRENORPHINE with FDV (Day 9) | 1110 (99.0)
  BUPRENORPHINE alone (Day 1) | 904 (109)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); BUPRENORPHINE(BUP) + Faldaprevir(FDV) on Day 9 vs. BUPRENORPHINE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.1915, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 108.36, 90% CI 2-sided [81.611 to 143.883], Standard Deviation 38.1 — The standard deviation is actually the intra-individual geometric coefficient of variation

11. Secondary Outcome: Pharmacodynamic Assessment of Withdrawal From Either Methadone or Buprenorphine/Naloxone Using the Subjective Opiate Withdrawal Scale (SOWS)-Change From Baseline
Description: The SOWS is a subjective scale self-evaluated by the subject. The SOWS shows items reflecting the common motor, autonomic, gastrointestinal, musculo-skeletal, and psychic symptoms of opiate withdrawal. Subjects are instructed to rate each symptom on a scale of 0 to 4 (0=not at all, 1=a little, 2=moderately, 3=quite a bit, 4=extremely) at designated times [c.f. Section 3.1]. The minimum possible SOWS score is 0, the maximum 64. The following subjective criteria are answered by the subject using the scale below: 1) I feel anxious, 2) I feel like yawning 3) I am perspiring, 4) My eyes are watering, 5) My nose is running, 6) I have goose flesh, 7) I am shaking 8) I have hot flushes, 9) I have cold flushes, 10) My bones and muscles ache, 11) I feel restless, 12) I feel nauseous, 13) I feel like vomiting, 14) My muscles twitch, 15) I have cramps in my stomach, 16) I feel like shooting up now. Higher score indicates increasing severity of opiate withdrawal syndrome.
Time Frame: Baseline, Day 2, Day 3, Day 4, Day 5, Day 6, Day 7, Day 8, Day 9, Day 10, Day 11, Day 12 and End of treatment
Population: This set included all subjects who took at least one dose of study drug.
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Methadone Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 15 | 19
units on a scale
  Day 2 | 0.0 [-4 to 2] | -1.0 [-11 to 2]
  Day 3 | 0.0 [-1 to 2] | 0.0 [-16 to 9]
  Day 4 (N=15,18) | 0.0 [-2 to 1] | 0.0 [-17 to 3]
  Day 5 (N=15,18) | 0.0 [-4 to 1] | -0.5 [-21 to 3]
  Day 6 (N=15,18) | 0.0 [-3 to 1] | -0.5 [-23 to 2]
  Day 7 (N=15,15) | 0.0 [-2 to 1] | -1.0 [-22 to 4]
  Day 8 (N=15,15) | 0.0 [-3 to 1] | -1.0 [-24 to 3]
  Day 9 (N=15,15) | 0.0 [-4 to 1] | -1.0 [-21 to 13]
  Day 10 (N=15,15) | 0.0 [-4 to 1] | -1.0 [-19 to 4]
  Day 11 (N=15,15) | 0.0 [-4 to 1] | -1.0 [-23 to 4]
  Day 12 (N=15,15) | 0.0 [-4 to 1] | -1.0 [-27 to 4]
  End of Treatment (EOT) (N=14,16) | 0.0 [-4 to 1] | -1.0 [-20 to 3]
Statistical Analysis 1: Comparison: Methadone Group; Pearson correlation of trough concentrations of R-methadone and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.04783, 95% CI 2-sided [-0.132750 to 0.224946]
Statistical Analysis 2: Comparison: Methadone Group; Pearson correlation of change from baseline for trough concentrations of R-methadone and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.39865, 95% CI 2-sided [-0.547072 to -0.222288]
Statistical Analysis 3: Comparison: Methadone Group; Pearson correlation of trough concentrations of S-methadone and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.11175, 95% CI 2-sided [-0.069336 to 0.284848]
Statistical Analysis 4: Comparison: Methadone Group; Pearson correlation of change from baseline for trough concentrations of S-methadone and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.16815, 95% CI 2-sided [-0.347870 to 0.025107]
Statistical Analysis 5: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of trough concentrations of Buprenorphine and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.01260, 95% CI 2-sided [-0.170160 to 0.194417]
Statistical Analysis 6: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of change from baseline for trough concentrations of Buprenorphine and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.02352, 95% CI 2-sided [-0.253932 to 0.296960]
Statistical Analysis 7: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of trough concentrations of norbuprenorphine and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = -0.05787, 95% CI 2-sided [-0.243920 to 0.132819]
Statistical Analysis 8: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of change from baseline for trough concentrations of norbuprenorphine and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.04052, 95% CI 2-sided [-0.218159 to 0.293233]
Statistical Analysis 9: Comparison: Buprenorphine/Naloxone (Suboxone); Pearson correlation of trough concentrations of naloxone and SOWS; Test type: Superiority or Other; Pearson Correlation Coefficient = 0.92231 — Confidence interval is not provided due to sparse data. There was only 1 patient for this analysis

12. Primary Outcome: Norbuprenorphine: Geometric Mean Steady-state AUC0-24 on Day 1 and on Day 9.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg*h/ml]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 12
[pg*h/ml]
  NORBUPRENORPHINE with FDV (Day 9) | 59200 (93.5)
  NORBUPRENORPHINE alone (Day 1) | 42900 (135)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); NORBUPRENORPHINE(BUP) + Faldaprevir(FDV) on Day 9 vs. NORBUPRENORPHINE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.6889, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 138.00, 90% CI 2-sided [97.20 to 195.92], Standard Deviation 50.7 — The standard deviation is actually the intra-individual geometric coefficient of variation

13. Primary Outcome: Norbuprenorphine: Geometric Mean Steady-state Cmax on Day 1 and on Day 9.
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg/mL]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 12
[pg/mL]
  NORBUPRENORPHINE with FDV (Day 9) | 3690 (91.9)
  NORBUPRENORPHINE alone (Day 1) | 2770 (126)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); NORBUPRENORPHINE(BUP) + Faldaprevir(FDV) on Day 9 vs. NORBUPRENORPHINE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.6188, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 132.86, 90% CI 2-sided [93.32 to 189.16], Standard Deviation 51.1 — The standard deviation is actually the intra-individual geometric coefficient of variation

14. Primary Outcome: Norbuprenorphine: Geometric Mean Steady-state C24hr on Day 1 and on Day 9.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg/mL]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 11
[pg/mL]
  NORBUPRENORPHINE with FDV (Day 9) | 2080 (102)
  NORBUPRENORPHINE alone (Day 1) | 2010 (113)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); NORBUPRENORPHINE(BUP) + Faldaprevir(FDV) on Day 9 vs. NORBUPRENORPHINE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.3152, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 112.03, 90% CI 2-sided [74.85 to 167.67], Standard Deviation 52.5 — The standard deviation is actually the intra-individual geometric coefficient of variation

15. Primary Outcome: Naloxone: Geometric Mean Steady-state AUC0-24 on Day 1 and on Day 9.
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg*h/ml]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 13
[pg*h/ml]
  NALOXONE with FDV (Day 9) | 971 (69.8)
  NALOXONE alone (Day 1) N=12 | 1000 (87.9)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); NALOXONE(BUP) + Faldaprevir(FDV) on Day 9 vs. NALOXONE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0107, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 98.94, 90% CI 2-sided [85.810 to 114.076], Standard Deviation 19.6 — The standard deviation is actually the intra-individual geometric coefficient of variation

16. Primary Outcome: Naloxone: Geometric Mean Steady-state Cmax on Day 1 and on Day 9.
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg/mL]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 14
[pg/mL]
  NALOXONE with FDV (Day 9) | 284 (107)
  NALOXONE alone (Day 1) N=13 | 357 (82.9)
Statistical Analysis 1: Comparison: Buprenorphine/Naloxone (Suboxone); NALOXONE(BUP) + Faldaprevir(FDV) on Day 9 vs. NALOXONE(BUP) alone on Day 1; Test type: Non-Inferiority or Equivalence — No formal testing, investigation of relative bioavailability; p = 0.0738, ANOVA — p-value for ratio outside interval 80% to 125%; [statistical method as in outcome 1, analysis 1]; Geometric mean ratio (%) = 94.33, 90% CI 2-sided [78.017 to 114.054], Standard Deviation 27.6 — The standard deviation is actually the intra-individual geometric coefficient of variation

17. Primary Outcome: Naloxone: Geometric Mean Steady-state C24hr on Day 1 and on Day 9.
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: [pg/mL]
Arm/Group | Buprenorphine/Naloxone (Suboxone)
Number analyzed (Participants) | 1
[pg/mL]
  NALOXONE with FDV (Day 9) | 23.4 (NA) — There was insufficient data to produce an estimate for dispersion. There was only 1 patients for this endpoint.
  NALOXONE alone (Day 1) | 25.6 (NA) — There was insufficient data to produce an estimate for dispersion. There was only 1 patient for this endpoint.

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Methadone Group | Buprenorphine/Naloxone (Suboxone)
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/19
Other Adverse Events (participants affected / at risk) | 12/15 | 18/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methadone Group (N=15) | Buprenorphine/Naloxone (Suboxone) (N=19)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 2 | 0
Nausea (Gastrointestinal disorders) | 7 | 10
Vomiting (Gastrointestinal disorders) | 5 | 5
Fatigue (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 3 | 7
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 2 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights..